CLINICAL TRIAL: NCT00631579
Title: Open-label, Multicenter Study of Repeated Doses of SR29142 (Rasburicase) as a Uricolytic Therapy for Hyperuricemia in Adult Patients With Leukemia or Lymphoma.
Brief Title: Rasburicase as a Uricolytic Therapy for Hyperuricemia in Patients With Leukemia or Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARD5290
Record Dates: First submitted 2008-02-26; First posted 2008-03-07 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: Hyperuricemia; Leukemia; Lymphoma
MeSH Terms: conditions — Hyperuricemia; Leukemia; Lymphoma | interventions — rasburicase; Urate Oxidase

INTERVENTIONS:
Drug: Rasburicase (SR29142)

SUMMARY:
The primary objectives of the study are to evaluate the safety and the efficacy in patients with malignant lymphoma or acute leukemia who are repeatedly administered for SR29142 5 days in two dosage groups.

Secondary objectives are to determine the pharmacokinetic (PK) parameters of SR29142 , to assess anti-SR29142 antibody production in patients with malignant lymphoma and acute leukemia, and to estimate the optimal dosage of SR29142 for Japanese patients from the results of efficacy and safety evaluations.

ELIGIBILITY:
Inclusion Criteria:

Patient suffering from:

* acute leukemia with white blood cell (WBC) count≥ 20,000/mm3 without regard to uric acid level ; or
* lymphoma,Stage ≥ III without regard to uric acid level; or
* lymphomas, Stage II with bulky disease; or
* lymphoma or leukemia, without regard to classification or morphology, with uric acid level ≥ 8.0 mg/dL, and lactate dehydrogenase (LDH) level ≥ twice the upper limit of normal (ULN).

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-04; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Safety via physical examination, laboratory tests and adverse events. Efficacy via plasma uric acid levels.

SECONDARY OUTCOMES:
Pharmacokinetic parameters and anti-SR29142 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: K.K., Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Tokyo, Japan

REFERENCES:
- [Derived] Ishizawa K, Ogura M, Hamaguchi M, Hotta T, Ohnishi K, Sasaki T, Sakamaki H, Yokoyama H, Harigae H, Morishima Y. Safety and efficacy of rasburicase (SR29142) in a Japanese phase II study. Cancer Sci. 2009 Feb;100(2):357-62. doi: 10.1111/j.1349-7006.2008.01047.x. PMID 19076979